CLINICAL TRIAL: NCT01112085
Title: Phase 2 Study of Microdoses of Ranibizumab in Diabetic Macular Edema - the MINIMA 2 Study
Brief Title: MIcrodoses of raNIbizumab in Diabetic MAcular Edema (MINIMA-2)
Acronym: MINIMA-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Especialistas en Retina Medica y Quirurgica Grupo de Investigacion (Network)
Collaborators: Centro de Retina Medica y Quirurgica S.C. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MINIMA-2
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema; Ranibizumab
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab 0.05mg (Experimental): Intravitreal injections of 0.05mg ranibizumab over 6 months then additional treatment with ranibizumab 0.05mg as needed (according to re-treatment criteria)
  Interventions: Drug: Ranibizumab 0.05mg
- Ranibizumab 0.5mg (Experimental): Intravitreal injections of 0.5mg ranibizumab over 6 months then additional treatment with ranibizumab 0.5mg as needed (according to re-treatment criteria)
  Interventions: Drug: Ranibizumab 0.5mg

INTERVENTIONS:
Drug: Ranibizumab 0.05mg — Intravitreal injections of 0.05mg ranibizumab over 6 months then additional treatment with ranibizumab 0.05mg as needed (according to re-treatment criteria)
  Arms: Ranibizumab 0.05mg
Drug: Ranibizumab 0.5mg — Intravitreal injections of 0.5mg ranibizumab over 6 months then additional treatment with ranibizumab 0.5mg as needed (according to re-treatment criteria)
  Arms: Ranibizumab 0.5mg

SUMMARY:
The objective of this study is to investigate if the drug ranibizumab administrated by microdose injection into the eye is safe and effective to treat diabetic macular edema.

DETAILED DESCRIPTION:
The MINIMA-2 Study is a multi-center clinical trial that initiated in order to investigate the effect of microdoses of ranibizumab in diabetic macular edema. The duration of the study is up to 13 months. Patients with diabetic macular edema will be randomized into 2 different groups. Consented subjects will receive monthly injections over a 6-month treatment period, and a 6 month follow-up and treatment period. Several eye examinations and procedures will be performed to evaluate response to the treatment. These include best corrected visual acuity testing (ETDRS), contrast sensitivity testing, ophthalmic examination, fluorescein angiography (FA)and macular thickness measurements based on optical coherence tomography (OCT). Serum chemistry, hematology and glycosylated hemoglobin HbA1c testing, urinalysis and pregnancy testing will be performed at screening visit (Days -14 to 0) and two more times during the study.

Approximately 72 patients with a baseline central foveal thickness by OCT of at least 270 will be included. The BCVA must be worst than 20/40 but better than or equal to 20/320 due diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older
* Subjects with diagnosis of diabetes mellitus (Type I or II)
* Signed informed consent
* Patient must be able to comply with study assessments
* Clinical sings and angiographic evidence of diabetic macular edema
* Central foveal thickness of at least 270 assessed by OCT
* Best corrected visual acuity of 20/40 to 20/320 (ETDRS chart) in the study eye

Exclusion Criteria:

* Patients who do not fulfill the inclusion criteria
* Use of any intraocular or periocular drug injection over the previous 3 months
* Macular or panretinal photocoagulation within 3 months of the study entry in the study eye
* High myopia (more than 6D)
* Any ocular disorders in the study eye that may confound interpretation of study results including patients with choroidal neovascularization, macular hole, retinal detachment, epiretinal membrane, ischemic maculopathy or any other retinal vascular disease such as vascular occlusive diseases.
* Vitreomacular traction
* Subretinal fibrosis
* Uncontrolled or advanced glaucoma
* Active ocular inflammation or history of active intraocular inflammation during the 6 months prior to enrollment of the study
* Any ophthalmic surgery performed within 3 months prior to study entry in the study eye
* Previous pars plana vitrectomy in the study eye
* History of ocular trauma of any type in the study eye
* Subjects with media opacities or abnormalities that would preclude observation of the retina in the study eye, per the investigator's judgement
* History of fluorescein allergy
* Known hypersensitivity to ranibizumab
* History of stroke or Myocardial infraction within 6 months
* Pregnancy, lactation or any women with no adequate contraception
* Participation in another simultaneous medical investigation or trial
* Any other condition that, in the opinion of the investigator, would produce a significant hazard or jeopardize the safety of the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 12 months
  Improvement in vision of best corrected visual acuity of 15 or more letters, or a final vision of 20/25 (50 letters) or better if best corrected visual acuity (BCVA) was 20/40 (40 letters)

SECONDARY OUTCOMES:
Mean change in central retinal thickness and volume by OCT | 6 months and 12 months
  Changes in central retinal thickness and volume assessed by optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Santos, MD PhD, Principal Investigator — Centro de Retina Médica y Quirúrgica S. C.
Locations (6):
- Centro Privado de Ojos Rogamosa SA y Fundación VER, Córdoba, Argentina
- Mexico (5):
  - Hospital San José, Guadalajara, Jalisco
  - Centro de Retina Médica y Quirúrgica S. C., Zapopan, Jalisco
  - Hospital Regional Valentín Gómez Farías, Zapopan, Jalisco
  - Hospital Universitario Doctor José Eleuterio González, Monterrey, Nuevo León
  - Hospital Central, San Luis Potosí City, San Luis Potosí